CLINICAL TRIAL: NCT02480881
Title: Effect of BMS-663068 on the Pharmacokinetics of a Combined Oral Contraceptive Containing Ethinyl Estradiol and Norethindrone Acetate in Healthy Female Subjects
Brief Title: A Drug-drug Interaction Study Between BMS-663068 and Oral Contraceptives in Healthy Female Volunteers (DDI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206279; AI438-019 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2015-06-18; First posted 2015-06-25 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Sequence A, B, C, and D (Experimental): Treatment A/Cycle 1: OC containing EE and progestin taken by mouth. Treatment B/Cycle 2: OC containing EE and progestin taken by mouth. Treatment C/Cycle 3: Loestrin 1.5/30 taken by mouth. Treatment D/Cycle 4: Loestrin 1.5/30 (alone) and Loestrin 1.5/30 with BMS-663068 taken by mouth.
  Interventions: Drug: BMS-663068; Drug: Oral Contraceptive; Drug: Loestrin 1.5/30

INTERVENTIONS:
Drug: BMS-663068 — Investigational product
Drug: Oral Contraceptive — Subject's existing combination OC tablet containing EE and progestin
Drug: Loestrin 1.5/30 — OC containing EE and norethindrone acetate (NEA)
  Other Names: Junel; Microgestin 1.5/30

SUMMARY:
This is an open-label, single sequence, 4-cycle, 4-treatment, drug-drug interaction (DDI) study in healthy female subjects on oral contraceptives (OC). There is no formal research hypothesis to be statistically tested. It is expected that coadministration of BMS-663068 with OC will not affect the pharmacokinetics (PK) of either ethinyl estradiol (EE) or norethindrone (NE).

ELIGIBILITY:
Inclusion Criteria:

* Healthy female nonsmoking subjects, ages 18 to 40 years, inclusive with a body mass index of 18.0 kg/m2 to 32.0 kg/m2, inclusive
* Women of child bearing potential with intact ovarian function by medical history and history of regular menstrual cycles must have been on a stable regimen of combination oral contraceptives containing EE and progestin (28 day regimen) without evidence of breakthrough bleeding or spotting for at least 2 consecutive months prior to Day -1

Exclusion Criteria:

* Any significant acute or chronic medical illness

Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2016-01-11 (Actual); Study Completion 2016-01-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter Cmax | From Day 21 of Treatment C/Cycle 3 to Day 21 of Treatment D/Cycle 4
  Pharmacokinetic parameter includes:
  maximal observed concentration (Cmax) for EE and NE.
Pharmacokinetic parameter AUC TAU | From Day 21 of Treatment C/Cycle 3 to Day 21 of Treatment D/Cycle 4
  Pharmacokinetic parameter includes:
  area under the concentration-time curve in one dosing interval (AUC(TAU)) for EE and NE.

SECONDARY OUTCOMES:
Clinical Safety as Measured by Adverse Event Monitoring. | From Day 1 (Treatment A/Cycle 1) to Day 22 (Treament D/Cycle 4)
  Adverse event monitoring
Clinical Safety as Measured by the Collection of Vital Signs. | From Day 1 (Treatment A/Cycle 1) to Day 22 (Treament D/Cycle 4)
  Vital signs assessments
Clinical Safety as Measured by the Collection of Electrocardiograms (ECGs). | From Day 1 (Treatment A/Cycle 1) to Day 22 (Treament D/Cycle 4)
  12-lead ECGs
Clinical Safety as measured by Physical Examination. | From Day 1 (Treatment A/Cycle 1) to Day 22 (Treament D/Cycle 4)
  Physical examinations
Clinical Safety as Measured by Clinical Laboratory Evaluations. | From Day 1 (Treatment A/Cycle 1) to Day 22 (Treament D/Cycle 4)
  clinical chemistry, hematology, and urinalysis.
Pharmacokinetic Parameter | From Day 21 of Treatment C/Cycle 3 to Day 21 of Treatment D/Cycle 4
  Pharmacokinetic parameter:
  -time of maximum observed concentration (Tmax) for EE and NE.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (2):
- United States (2):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, San Antonio, Texas